CLINICAL TRIAL: NCT02614911
Title: Host-Microbiota Interactions Across the Gut Immune System: Characterization of Phenotype and Genotype of Early Onset Enteropathies
Brief Title: Characterization of Phenotype and Genotype of Early Onset Enteropathies
Acronym: IMMUNOBIOTA
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IMIS2014-01
Record Dates: First submitted 2015-11-10; First posted 2015-11-25 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Disease
Keywords: Early Onset Entheropathy
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of:
  * blood samples
  * feces
  * biopsies (intestine / skin)
  * saliva
  * urina
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sick patients: Biological sampling of blood for all patients. Biological sampling of saliva, biopsies (skin and endoscopic), feces, for some patients
  Interventions: Other: Biological sampling
- Healthy relatives: Biological sampling of blood for all healthy relatives
  Interventions: Other: Biological sampling

INTERVENTIONS:
Other: Biological sampling — Biological sampling including blood, feces, biopsies...

SUMMARY:
This study has been set up in order to characterize phenotypes and genotypes of patients with early onset enteropathies.

In that goal, Investigators will collect biological samples (mainly blood) of patients suffering from early onset enteropathies and their healthy relatives.

DETAILED DESCRIPTION:
This study specifically aims at the genetic analysis of early onset enteropathies with the goal in mind to delineate human pathways necessary to maintain intestinal homeostasis despite the considerable density of microbes colonizing the distal part of the human intestine.

ELIGIBILITY:
Main Inclusion Criteria:

* Severe chronic enteropathy
* Patients developing their first symptoms within the first 6 years of life and, in priority within the first two years of life, or patients with a disease of later onset, in case of a familial history suggestive of inherited mutations notably in families comprising several affected members
* OR : Be a patient's relative, even if presenting with enteropathy of later onset.

Main Exclusion Criteria:

* Subject having participated to any therapeutical clinical study in the 30 days preceding the inclusion in this study,

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion of patients with chronic severe entheropathy and of their healthy relatives
Sampling Method: Probability Sample
Enrollment: 1445 (Estimated)
Dates: Start 2014-06-16 (Actual); Primary Completion 2054-06-15 (Estimated); Study Completion 2054-06-15 (Estimated)

PRIMARY OUTCOMES:
Increasing the current rate (20%) of genetic characterization of early onset entheropathies | 40 years
  Currently, around 20% of early onset entheropathies are genetically characterized. Investigators want to increase this rate via this research protocol.
  Our long term objective is to characterize phenotypes and genotypes of patients with early onset enteropathies.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ruemmele, Principal Investigator — Necker - Enfants Malades Hospital
Locations (12):
- France (12):
  - Centre Hospitalier Pellegrin-Enfants, Bordeaux
  - Hôpital pédiatrique de Lyon, Bron
  - Hôpital Jeanne de Flandre, CHRU de Lille, Lille
  - Hôpital d'enfants de la Timone, Marseille
  - Hôpital Saint Antoine, Paris
  - Necker - Enfants Malades Hospital, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Trousseau, Paris
  - Hôpital Sud, Rennes
  - CHU Hautepierre, Strasbourg
  - Hôpital des Enfants, Toulouse
  - Hôpital Clocheville, CHU de Tours, Tours